CLINICAL TRIAL: NCT01049165
Title: Placebo-Controlled, Ascending Single-Dose Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of BMS-813160 in Healthy Subjects
Brief Title: Single Ascending Dose (BMS-813160) Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: CV202-001
Record Dates: First submitted 2010-01-12; First posted 2010-01-14 (Estimated); Last update posted 2011-02-11 (Estimated); Status verified 2011-02

CONDITIONS: Accelerated Intimal Hyperplasia
MeSH Terms: interventions — BMS-813160

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (9):
- Arm 1 (BMS-813160 or placebo) (Active Comparator)
  Interventions: Drug: BMS-813160; Drug: Placebo
- Arm 2 (BMS-813160 or placebo) (Active Comparator)
  Interventions: Drug: BMS-813160; Drug: Placebo
- Arm 3 (BMS-813160 or placebo) (Active Comparator)
  Interventions: Drug: BMS-813160; Drug: Placebo
- Arm 4 (BMS-813160 or placebo) (Active Comparator)
  Interventions: Drug: BMS-813160; Drug: Placebo
- Arm 5 (BMS-813160 or placebo) (Active Comparator)
  Interventions: Drug: BMS-813160; Drug: Placebo
- Arm 6 (BMS-813160 or placebo) (Active Comparator)
  Interventions: Drug: BMS-813160; Drug: Placebo
- Arm 7 [14C] BMS-813160 (Active Comparator)
  Interventions: Drug: [14C] BMS-813160
- Arm 8 (BMS-813160 or placebo) (Active Comparator)
  Interventions: Drug: Placebo; Drug: BMS-813160
- Arm 9 (BMS-813160 or placebo) (Active Comparator)
  Interventions: Drug: BMS-813160

INTERVENTIONS:
Drug: BMS-813160 — Oral Solution, Oral, 5 mg, Single dose, 1 day
  Arms: Arm 1 (BMS-813160 or placebo)
Drug: BMS-813160 — Oral Solution, Oral, 20 mg, Single dose, 1 day
  Arms: Arm 2 (BMS-813160 or placebo)
Drug: BMS-813160 — Oral Solution, Oral, 60 mg, Single dose, 1 day
  Arms: Arm 3 (BMS-813160 or placebo)
Drug: BMS-813160 — Oral Solution, Oral, 150 mg, Single dose, 1 day
  Arms: Arm 4 (BMS-813160 or placebo)
Drug: BMS-813160 — Oral Solution, Oral, 300 mg, Single dose, 1 day
  Arms: Arm 5 (BMS-813160 or placebo)
Drug: BMS-813160 — Oral Solution, Oral, 600 mg, Single Dose, 1 day
  Arms: Arm 6 (BMS-813160 or placebo)
Drug: [14C] BMS-813160 — Oral Solution, Oral, 150 mg, Single Dose, 1 day
  Arms: Arm 7 [14C] BMS-813160
Drug: Placebo — Oral Solution, Oral, 0 mg, Single Dose, 1 day
  Arms: Arm 1 (BMS-813160 or placebo); Arm 2 (BMS-813160 or placebo); Arm 3 (BMS-813160 or placebo); Arm 4 (BMS-813160 or placebo); Arm 5 (BMS-813160 or placebo); Arm 6 (BMS-813160 or placebo); Arm 8 (BMS-813160 or placebo)
Drug: BMS-813160 — Oral Solution, Oral, 1200 mg, Single dose, 1 day
  Arms: Arm 8 (BMS-813160 or placebo)
Drug: BMS-813160 — Oral Solution, Oral, 2000 mg, Single Dose, 1 day
  Arms: Arm 9 (BMS-813160 or placebo)

SUMMARY:
The primary purpose of this study is to evaluate the safety and tolerability of single oral doses of BMS-813160 in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Men and women (not of child bearing potential) ages 18 to 45
* Healthy subjects as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs, and clinical laboratory determinations

Exclusion Criteria:

* Women of Child Bearing Potential
* Organ dysfunction or any clinically significant deviation from normal in medical history, physical examination, ECGs, and clinical laboratory determinations

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2010-02; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Safety will be assessed by clinical laboratory results, ECGs, vital signs, and reported adverse events | Dosing through Day 5

SECONDARY OUTCOMES:
Pharmacokinetics of BMS-813160 | 9 times after dosing
Pharmacodynamics (Plasma MCP-1) | 9 times post dose
Pharmacodynamics (Circulating monocytes) | 5 times post dose
Pharmacodynamics (CCR5 phosphorylation and internalization in whole blood) | 5 times post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Covance Clinical Research Unit, Inc., Madison, Wisconsin, United States

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx